CLINICAL TRIAL: NCT01310855
Title: Multi-Center, Randomized, Double-Blind Phase II Study Comparing Cediranib (AZD2171) Plus Gefitinib (Iressa, ZD1839) With Cediranib Plus Placebo in Subjects With Recurrent/Progressive Glioblastoma (DORIC Trial)
Brief Title: Cediranib Maleate With or Without Gefitinib in Treating Patients With Recurrent or Progressive Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed to recruitment early due to AstraZeneca not developing cediranib further
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000696313; UCL-10/0035; ZENECA-ISSRECE00002; EUDRACT-2010-021531-13; CRUKE/10/044
Record Dates: First submitted 2011-03-05; First posted 2011-03-09 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Glioblastoma
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — cediranib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cediranib & Gefitinib (Active Comparator): Cediranib maleate 30mg od orally and gefitinib 500mg od orally. Each cycle of treatment lasts 6 weeks. Treatment will continue until confirmation of progression, patient decision or the development of unacceptable toxicity (if there is radiological progression only treatment can continue if the investigator has the opinion that the patient is receiving benefit.
  Interventions: Drug: cediranib maleate; Drug: gefitinib
- Cediranbib & placebo (Placebo Comparator): Cediranib maleate 30mg od orally and placebo 500mg od orally. Each cycle of treatment lasts 6 weeks. Treatment will continue until confirmation of progression, patient decision or the development of unacceptable toxicity (if there is radiological progression only treatment can continue if the investigator has the opinion that the patient is receiving benefit.
  Interventions: Drug: cediranib maleate; Drug: Placebo

INTERVENTIONS:
Drug: cediranib maleate
Drug: gefitinib
  Arms: Cediranib & Gefitinib
Drug: Placebo
  Arms: Cediranbib & placebo

SUMMARY:
RATIONALE: Cediranib Maleate and gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether cediranib maleate given together with gefitinib is more effective than cediranib maleate given alone in treating patients with recurrent or progressive glioblastoma.

PURPOSE: This randomized phase II trial is studying the side effects of giving cediranib maleate together with gefitinib and to see how well it works compared with giving cediranib maleate together with a placebo in treating patients with recurrent or progressive glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare progression-free survival, overall survival, radiological response, and safety and tolerability of cediranib maleate in combination with gefitinib versus cediranib maleate in combination with a placebo in patients with recurrent or progressive glioblastoma following standard front-line treatment.

OUTLINE: This is a multicenter study.

Patients receive cediranib maleate and gefitinib or cediranib maleate and a placebo once daily on days 1-42. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected from some patients for genetic profiling and biomarker analysis.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed glioblastoma
* Measurable disease by MRI
* Completed standard first-line treatment for glioblastoma including surgery (unless not received due to anatomical location), radiotherapy and temozolomide (last dose given at least 28 days prior to enrollment)

  * No other prior treatment for glioblastoma except Gliadel or steroids
* Recurrent or progressive disease after standard first-line treatment

  * No disease progression within 3 months of completion of radiotherapy
* No intra- or peri-tumoral hemorrhage

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Mini-mental status score ≥ 15
* Life expectancy ≥ 12 weeks
* Serum bilirubin, ALT/AST, creatinine, and urine protein normal
* Adequate bone marrow reserve
* Not pregnant or nursing
* Normal ECG
* No history of familial long QT syndrome
* No absorption or swallowing difficulties
* No uncontrolled hypertension or cardiac ventricular arrhythmias
* No current or history of uncontrolled hypertension or requiring maximal doses of calcium channel blockers
* No severe or uncontrolled disease
* No history of lung disease
* No recent hemorrhage or hemoptysis
* No known hypersensitivity to cediranib maleate, gefitinib, or any excipients
* No history of other malignancies except adequately treated basal cell or squamous cell carcinoma or carcinoma in situ within the past 5 years, unless disease-free for 2 years with tissue diagnosis
* No known HIV positivity
* No known hepatitis B or C infection
* No unhealed surgical incision
* Not involved in planning or conducting this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior anticancer therapy, including radiotherapy
* At least 3 months since prior cranial radiation
* At least 30 days since prior investigational drugs
* At least 28 days since prior craniotomy
* At least 2 weeks since prior enzyme-inducing antiepileptic drugs
* At least 2 weeks since prior and no concurrent dexamethasone (> 8 mg/day) or equivalent
* At least 14 days since prior major surgery or brain biopsy
* No concurrent steroids OR on stable dose 5 days prior to baseline MRI
* No other concurrent anticancer therapy, except for steroids (dexamethasone only)
* No previous enrollment on the current study
* No prior inhibitors of angiogenesis, EGFR, or downstream targets
* No prior radiosurgery or brachytherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mulholland, PhD, MRCP, MSC, MBBS, Principal Investigator — University College London Hospitals
Locations (10):
- United Kingdom (10):
  - University College Hospital, London, England
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Royal Surrey County Hospital, Guildford
  - Castle Hill Hospital, Hull
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Brown N, McBain C, Nash S, Hopkins K, Sanghera P, Saran F, Phillips M, Dungey F, Clifton-Hadley L, Wanek K, Krell D, Jeffries S, Khan I, Smith P, Mulholland P. Multi-Center Randomized Phase II Study Comparing Cediranib plus Gefitinib with Cediranib plus Placebo in Subjects with Recurrent/Progressive Glioblastoma. PLoS One. 2016 May 27;11(5):e0156369. doi: 10.1371/journal.pone.0156369. eCollection 2016. PMID 27232884

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Trial closed prematurely because cediranib manufacture was discontinued by AZ. Only 38 patients were recruited
Groups:
- Cediranib & Gefitinib: Cediranib maleate 30mg od orally and gefitinib 500mg od orally. Each cycle of treatment lasts 6 weeks. Treatment will continue until confirmation of progression, patient decision or the development of unacceptable toxicity (if there is radiological progression only treatment can continue if the investigator has the opinion that the patient is receiving benefit.
  cediranib maleate
  gefitinib
- Cediranbib & Placebo: Cediranib maleate 30mg od orally and placebo 500mg od orally. Each cycle of treatment lasts 6 weeks. Treatment will continue until confirmation of progression, patient decision or the development of unacceptable toxicity (if there is radiological progression only treatment can continue if the investigator has the opinion that the patient is receiving benefit.
  cediranib maleate
  Placebo
Period: Overall Study
Arm/Group | Cediranib & Gefitinib | Cediranbib & Placebo
Started (112 patients were to be recruited but 38 recruited due to the early discontinuation of cediranib) | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib & Gefitinib | Cediranbib & Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 54.4 [30 to 71] | 56.9 [40 to 69] | 55.7 [30 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival (PFS) defined as the time from the date of randomisation to the date of first progression or death due to any cause, whichever one comes first.
  The progression definition will be based on modified RANO criteria (Wen 2010), such that progression will be defined as the earliest time that at least one of the following occurs:
  1. Clinical deterioration
  2. Failure to return for evaluation as a result of death or deteriorating condition
     Or, by retrospective radiographic central review:
  3. Any new lesion
  4. Increase in ≥25% of sum of the products of perpendicular diameters of enhancing lesions compared with baseline scan, on stable or increasing doses of steroids (dexamethasone) compared to baseline (T1 post-contrast scan)
  5. Clear progression of non-measureable disease
  6. Significant increase in T2/FLAIR non-enhancing lesion - on stable or increasing steroids (dexamethasone) compared with baseline or best response not caused by co-morbid events.
Time Frame: from the date of randomisation to the date of first progression or death due to any cause, until 6 months from the date the last patient finished trial treatment (the day after the date that the last trial drug was taken)
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cediranib & Gefitinib | Cediranbib & Placebo
Number analyzed (Participants) | 19 | 19
months | 3.6 [2.8 to 4.1] | 2.8 [2.1 to 3.4]

2. Secondary Outcome: Overall Survival
Time Frame: from date of randomization to date of Death due to any cause.
Reporting Status: Not Posted

3. Secondary Outcome: Radiographic Response Rate
Time Frame: from baseline scan to six week and 12 week scans
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free Survival Rate at 6 Months
Time Frame: from the date of randomisation to 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Steroid Use
Time Frame: from randomization to first increase in dexamethasone dose
Reporting Status: Not Posted

6. Secondary Outcome: Time to Deterioration of Neurological Status
Time Frame: from date of randomization to the date of first neurological status worsening in comparison to baseline (first of 2 confirmatory reports at 2 consecutive visits, 6 weeks apart) as assessed by the clinician, or until date of death, whichever is first.
Reporting Status: Not Posted

7. Secondary Outcome: Safety and Tolerability
Time Frame: from date of randomisation to death
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Cediranib & Gefitinib: Cediranib maleate 30mg od orally and gefitinib 500mg od orally. Each cycle of treatment lasts 6 weeks. Treatment will continue until confirmation of progression, patient decision or the development of unacceptable toxicity (if there is radiological progression only treatment can continue if the investigator has the opinion that the patient is receiving benefit.
  Due to the early discontinuation of Cediranib by AZ, the trial was discontinued early so that only 38 patients (19 per arm) were recruited. One patient in the Cediranib arm did not complete their patient diary, and it was not known how much of the trial treatment they had. Therefore the adverse events reported by the patient could not be attributed to the trial treatment and they were excluded from all analyses.
- Cediranbib & Placebo: Cediranib maleate 30mg od orally and placebo 500mg od orally. Each cycle of treatment lasts 6 weeks. Treatment will continue until confirmation of progression, patient decision or the development of unacceptable toxicity (if there is radiological progression only treatment can continue if the investigator has the opinion that the patient is receiving benefit.
  Due to the early discontinuation of Cediranib by AZ, the trial was discontinued early so that only 38 patients (19 per arm) were recruited.
Arm/Group | Cediranib & Gefitinib | Cediranbib & Placebo
Serious Adverse Events (participants affected / at risk) | 5/18 | 7/19
Other Adverse Events (participants affected / at risk) | 16/18 | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib & Gefitinib (N=18) | Cediranbib & Placebo (N=19)
Pulmonary embolism (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
dysphasia (Nervous system disorders) | 1 | 0
headache (Nervous system disorders) | 1 | 0
movement involuntary (Nervous system disorders) | 1 | 0
other, hemispatial neglect of right arm (Nervous system disorders) | 1 | 0
other - right arm numbness (Nervous system disorders) | 1 | 0
other - right homonymous hemiopia (Nervous system disorders) | 1 | 0
other - reduced mobility (Nervous system disorders) | 1 | 0
other - weakness in right arm (Nervous system disorders) | 1 | 0
seizure (Nervous system disorders) | 2 | 0
stroke (Nervous system disorders) | 1 | 0
confusion (Psychiatric disorders) | 1 | 0
other (Infections and infestations) | 0 | 1
lung infection (Infections and infestations) | 0 | 1
sepsis (Infections and infestations) | 2 | 0
skin infection (Infections and infestations) | 1 | 0
wound infection (Infections and infestations) | 1 | 0
cushingoid (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib & Gefitinib (N=18) | Cediranbib & Placebo (N=19)
hypertension (Vascular disorders) | 5 | 1
thromboembolic event (Vascular disorders) | 1 | 1
fatigue (General disorders) | 4 | 6
cognitive disburbance (Psychiatric disorders) | 2 | 0
confusion (Psychiatric disorders) | 1 | 0
fall (Injury, poisoning and procedural complications) | 0 | 2
lymphopenia (Investigations) | 3 | 2
alanine aminotransferase increased (Investigations) | 0 | 2
cholesterol high (Investigations) | 0 | 1
hypertrigylceridomia (Investigations) | 0 | 1
GGT increased (Investigations) | 0 | 1
haemorrage (Blood and lymphatic system disorders) | 0 | 1
dysphasia (Nervous system disorders) | 1 | 2
headache (Nervous system disorders) | 2 | 1
pain (Nervous system disorders) | 1 | 1
seizure (Nervous system disorders) | 1 | 0
other (Nervous system disorders) | 1 | 0
movements involuntary (Nervous system disorders) | 1 | 0
paresthesia (Nervous system disorders) | 1 | 0
eye disorder (Eye disorders) | 2 | 0
blurred vision (Eye disorders) | 1 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 0
mucositis oral (Gastrointestinal disorders) | 1 | 0
stomatitis (Gastrointestinal disorders) | 0 | 1
skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
muscle weakness right handed (Musculoskeletal and connective tissue disorders) | 1 | 0
generalised muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
cushingoid (Endocrine disorders) | 0 | 1
anorexia (Metabolism and nutrition disorders) | 1 | 3
hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
rash pustular (Infections and infestations) | 2 | 1
sepsis (Infections and infestations) | 2 | 0
infection (Infections and infestations) | 1 | 0
aspartate aminotransferase increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The excerpts below are present on all site agreements between site staff (including PI) and the sponsor:

* The Site shall ensure that only those of its employees or officers directly concerned with the conduct of the Trial at the Site shall have access to the Confidential Information relating to the Trial.
* The Site agrees it will not publish any information, data or results without the express written permission of the TMG, such permission not to be unreasonably withheld.